CLINICAL TRIAL: NCT06767241
Title: Subtle Pulse Electro-biological Recovery Apparatus (SPERA) for COVID-19 - a Proof of Concept Study
Brief Title: Transcranial Non-invasive Electrical Stimulation of the Vagus Nerve in Hospitalized Moderate-to-severe COVID-19 Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Medicine and Pharmacy "Victor Babes" Timisoara (Other)
Responsible Party: Principal Investigator, Basaraba Gabriela Lavinia, Center for Research and Innovation in Precision Medicine of Respiratory Diseases, Department of Pulmonology, University of Medicine and Pharmacy Timisoara, University of Medicine and Pharmacy "Victor Babes" Timisoara
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 10669/14.12.2020
Record Dates: First submitted 2024-12-05; First posted 2025-01-09 (Actual); Last update posted 2025-01-09 (Actual); Status verified 2024-12

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Non-invasive auricular vagus nerve stimulation (Active Comparator): Transcranial electrical stimulation of the vagus nerve delivered through the SPERA device on top of the standard care treatment
  Interventions: Device: Non-invasive auricular vagus nerve stimulation; Other: Standard Medical Therapy
- Control group (Placebo Comparator): Standard of care treatment
  Interventions: Other: Standard Medical Therapy

INTERVENTIONS:
Device: Non-invasive auricular vagus nerve stimulation — Non-invasive transcranial direct current auricular vagus nerve stimulation (tDC-aVNS)
  Arms: Non-invasive auricular vagus nerve stimulation
Other: Standard Medical Therapy — Standard of care treatment for moderate to severe COVID-19

SUMMARY:
Subtle Pulse Electro-biological Recovery Apparatus (SPERA) is an innovative device which delivers digital subliminal pulse stimulation trans cranially to auricular branches of the central nervous system and modulates the anti-inflammatory reflexes mediated by afferent and efferent fibers of the Vagus Nerve. The aim of this single center, interventional study was to assess the efficacy and safety of non-invasive trans-cranial Direct Current auricular Vagus Nerve Stimulation (aVNS) delivered by SPERA in the resolution of inflammatory insults in patients with SARS-CoV-2 infection. Patients hospitalized with moderate-to-severe COVID-19 will be enrolled in the study. Inclusion criteria: RT-PCR confirmed SARS-CoV-2 infection, lung involvement as demonstrated by chest CT scan, increased risk for cytokine storm (CRP>46mg/L, ferritin>250ng/mL). Key exclusion criteria: critical patients upon admission, requiring ICU care. SPERA therapy will be administered on top of the standard of care treatment for consecutive patients satisfying the above mentioned criteria.

DETAILED DESCRIPTION:
Can non-invasive transcranial Direct Current Auricular Vagus Nerve Stimulation (tDC-aVNS) inhibit Cellular and Systemic Inflammation in COVID-19, reducing risk of longer hospitalization, chronic morbidity and mortality?

A clinical research protocol to determine if non-invasive trans-cranial Direct Current auricular Vagus Nerve Stimulation (tDC-aVNS) decreases pro-inflammatory Cytokines and Chemokines in COVID-19: a Proof of Concept Trial of adults with moderate to severe symptomology, at greatest danger of SARS-Cov2 Cytokine Storm.

Objectives:

To observe how many patients with moderate-severe forms of Covid-19 will need to be admitted to the ICU with hyper-inflammation (Cytokine Storm) after application of Subtle Pulse Electro-biological Recovery Apparatus (SPERA) in addition to the Standard of Care (SOC), comparing tDC-aVNS from Prescription group and a Control group who receive only SOC.

SOC observations for all patients will include: a CT scan prior to admission or in the first days after admission. Blood samples collected for hemoleucogram with FBC, coagulation parameters, D-dimers, fibrinogen, CRP, procalcitonin, LDH, ferritin, ALT, AST, urea, creatinine, glucose, sodium, potassium, GGT, bilirubin. The clinical status (symptoms and clinical signs) will be checked daily and the vital signs: BP, pulse rate, temperature, oxygen saturation will also be measured regularly. An ECG will be routinely performed and cardiologist's advice will be sought on anticoagulation treatment. Additional investigations will be performed upon request as needed (such as inflammatory cytokines, etc). Further objective measures will include: time to clinical recovery, clinical status, hospital length of stay, number of days with supplemental oxygen and/or non-invasive ventilation, mortality rate.

Introduction:

The primary challenge in hospital wards treating patients with SARS-Cov-2 is to identify safe and effective therapies to prevent or resolve cellular and systemic inflammation caused by this novel virus without compromising protective innate autoimmune responses. Those with severe infection are at high risk of acute complications, intractable new co-morbidities and lengthy hospitalization. Physicians struggle to resolve pulmonary inflammation before occurrence of Acute Respiratory Distress Syndrome (ARDS). Patients can progress rapidly to the devastating hyper-inflammatory response and tissue damage known as Cytokine Storm (CS) with coagulation, multi-organ failure and greatest danger of mortality. Avoiding this conclusion and restoring homeostasis presents a double-edged sword if pharmacology for inhibiting inflammation also compromises the innate immune system. Therefore, the investigators will conduct an open label, interventional, proof of concept clinical trial to assess the safety and effectiveness of non-invasive, subliminal amperage, auricular Vagus Nerve stimulation (aVNS), of the adult human anti-inflammatory pathways in hospitalized patients with moderate-severe Covid-19.

SPERA delivers digital subliminal pulse stimulation transcranially (tDCS) to auricular branches of the Central Nervous System (CNS), it is claimed, by modulating afferent and efferent fibres of the Vagus Nerve (VN). Murine and human studies have demonstrated the efficacy and safety of vagus nerve stimulation (VNS) in the resolution of inflammatory insults including sepsis. Surgically implanted electrodes have hitherto been employed to overcome impedance of skin and bone to deliver therapeutic pulse frequencies to VN. SPERA however, employs a non-invasive auricular access to the vagal afferent - efferent feedback loop, which moderates and mediates homeostasis and inflammation from brain throughout the body.

Methods and materials:

To identify patients with comparably moderate-severe expression of COVID-19 we will adopt criteria set out in Table 4 of the Carricchio predictive model (Caricchio R, et al. Preliminary predictive criteria for COVID-19 cytokine storm. Ann. Rheum Dis 2020; 0: 1-8.) Those patients who meet this criteria remain three times longer in hospital and suffer six times higher loss of life. Our early ability to predict which patients will most probably develop CS could help target inflammatory cytokine-inhibition strategies (including non-invasive aVNS), shorten hospitalization, reduce mortality and improve clinical outcomes.

The investigators will prioritize those most likely to develop COVID Cytokine Storm (COVID-CS) and requiring early therapeutic intervention to resolve acute immune system dysfunction. SARS-Cov2 associated CS is considered to be a unique form of a hyper-inflammatory response. Criteria classifying other forms of CS, Macrophage Activation Syndrome (MAS), Haemophagocytic Lymphohistiocytosis (HLH) and the HScore, does not sufficiently identify and predict COVID-CS. Therefore, patient selection for our clinical trial of SPERA will be made using the Caricchio predictive model identifying those at high risk of progressing to CS. Patients, fulfilling this triage criteria, present with symptoms comprising three clusters of laboratory analysis:

* Inflammation;
* Cell death and tissue damage;
* Prerenal electrolyte imbalance. These clusters accurately predict viral infection severity most likely to develop into CS in COVID-19, thereby raising the urgency of early intervention to inhibit pro-inflammatory damage and restore autoimmune dysfunction.

The investigators will consider patients with a positive RT-PCR test for COVID-19, having moderately-severe symptoms, expressed by extensive fatigue, confusion, abdominal and respiratory symptoms (according to the Caricchio severity criteria clusters 4-6, which demonstrate a sensitivity of 0.85 and a specificity of 0.8) and evidence of COVID-19 pneumonia on the chest CT scan among those hospitalized at "Victor Babes" Infectious Diseases and Pulmonology Clinical Hospital, Timisoara.

The patients agreeing to enrol in the study by signing the Informed Consent Form will receive a tDC-aVNS anti-inflammatory prescription by applying the SPERA device 4+4 hours each day, between 1 and 7 days, in addition to the standard of care. The control group will consist of hospitalized patients with COVID-19, matched by age, sex and severity of disease. In the study group we will differentiate at what time the SPERA aVNS anti-inflammatory prescription was applied following onset of symptoms (first, second week of infection).

A total of 30 male and female adults with moderate-severe Covid-19 symptomology will be enrolled to receive the SPERA anti-inflammatory digital prescription by trans-cranial Direct Current - auricular Vagus Nerve Stimulation in addition to the standard of care. All subjects will undergo an initial clinical evaluation including vital signs measurement and a blood draw between 07:30 and 9:30am, followed by stimulation at 10am-13.45pm, with tDC-aVNS Prescription. The SOC Control group will receive no SPERA digital stimulation, while patients in the tDC-aVNS prescription group will receive a second session of stimulation between 14:15pm -18.00pm. Additional blood samples will be drawn again 24 hours after the first stimulation session. Samples will be measured for inflammatory markers and pro-inflammatory cytokines (biomarker IL-6) using ELISA. Statistical comparative analyses within and between groups will be calculated.

Intervention:

All patients will receive the same clinical standard of care. The active treatment group will additionally receive SPERA aVNS, a digital anti-inflammatory prescription group. The SPERA device will produce a subliminal low amperage, low-voltage electrical square wave pulse with zero-charge component (at pre-programmed frequencies-Hz, variable wavelengths-milliseconds and pulse trains/pauses). Upon auricular Cymba Conchae (CC) montage application of the device, it will generate subtle pulses at a maximum output of 10V and subliminal 10-12 microAmp current, delivering a pre-programmed digital inflammation-inhibiting prescription (10 volunteers), or sham stimulation (10 volunteers), the Control SOC group will receive no aVNS stimulation (10 volunteers). Anod/Cathode ionized carbon or metallic auricular ear-clip electrodes applied by the research team will enable delivery of auricular digital vagus nerve stimulation. In the tDC-aVNS prescription group the investigation team will place the device electrodes on the ears at the CC designated point of stimulation. In the inflammation-inhibiting tDC-aVNS prescription group there will be no noticeable tingling or sensation of electrical pulse during the stimulation sessions. (SPERA) devices will be applied to right and left ears of the tDC-aVNS prescription group in the CC montage throughout the 4+4 hour aVNS stimulation sessions.

Research Design:

Hospitalised volunteers with moderate-severe COVID-19 will be recruited at the designated research facility for two sessions during two consecutive days. The Standard Operating Procedure (SOP) for SPERA COVID-19 Clinical Trials, with informed consent, will be rigorously applied by SPERA Trained Workers (STW). Patients from each group will undergo an initial blood draw DAY1 between 07:30 and 9:30am, followed by stimulation with tDC-aVNS Anti-inflammation digital Prescription (active treatment group); or no SPERA, just SOC (control group). Stimulation for tDC-aVNS Prescription group will last for four hours in the morning and four hours in the afternoon DAY1 from 10.00-13.45 and 14.15-18.00. The subjects will be examined again at the designated research facility the following morning. On DAY2, research staff will ascertain any changes to subject's medical history or adverse events, electrocardiographic findings, and vital signs and perform a physical examination. A second blood draw will be taken on DAY2, 24 hours after the first stimulation session. The primary endpoint of this study will be the time to recovery defined as the time to hospital discharge with or without home oxygen requirement. Secondary outcomes include the number of patients requiring admission to the ICU, hospital length of stay, number of days with supplemental oxygen and/or non-invasive ventilation, mortality rate and detection of percent change in inflammatory markers and pro-inflammatory cytokines (IL-6).

Hypothesized Results:

Signs of systemic inflammation will be prominent in the COVID-CS cohort, indicating significantly higher levels of ferritin, C-Reactive Protein (CRP), LDH and fibrinogen. CRP, an acute-phase reactant protein of hepatic origin, increases following interleukin-6 (IL-6) secretion by macrophages and T cells. Harmful inflammation will be confirmed by the elevation of IL-6 in most COVID-19 patients, but significantly higher (Caricchio et al. mean: 35 vs 96pg/mL) in COVID-CS. This clinical study will observe whether a significant percent decrease occurs following SPERA digital prescription in levels of inflammation; cell death and tissue damage; prerenal electrolyte imbalance; with the pro-inflammatory cytokine IL-6 as a biomarker. This clinical trial of tDC-aVNS will be conducted in hospitalized volunteers with moderate-severe COVID-19 infection. In mammalian studies of sepsis and VNS, levels of pro-inflammatory cytokines were inhibited, including IL-1b, IL-6, tumor necrosis factor alpha (TNFa) levels, and chemokine, interleukin IL-8, macrophage inflammatory protein [MIP]-1a, and monocyte chemo-attractant protein [MCP]-1. In SOC only group, if consistent with previous studies there might be a significant percent increase in pro-inflammatory biomarkers at 24 hours (p<0.05). At 24 hours, in the tCD-aVNS Prescription group, according to previous studies, might be observed to have a greater percent decrease in pro-inflammatory biomarker concentration (p<0.05) compared to SOC group. The tCD-aVNS prescription group, based on previous published VNS research, might have a greater percent decrease in inflammatory markers and pro-inflammatory cytokines at 24 hours (p<0.05) in comparison to SOC group.

Conclusions:

If SPERA non-invasive VNS down-regulates (inhibits) inflammatory cytokine release (IL-6, IL-1b, TNFa etc, analyzing IL-6 as primary biomarker) as hypothesized, it may be that non-invasive auricular tDCS of the VN could safely resolve and prevent CS risk in COVID-19. It is supposed that VNS restores dysfunctional afferent - efferent communication, which may be a cause of unregulated hyper-inflammatory insults. tDC-aVNS would be an inexpensive, novel and potentially ubiquitous treatment for cytotoxic cellular and systemic inflammation. This could be an adjunct or alternative to cytokine-neutralizing and anti-inflammation pharmacology, without unwelcome autoimmune system side-effects. Further clinical trials could extend this tool in prophylaxis, ICU, and chronic recovery stages of SARS-Cov2. If proven safe and effective, clinical benefits would be reduced morbidity and mortality; less time in hospital; quicker and more complete viral clearance. Moreover, it is possible that that on-going SPERA VNS prescription research, applied to COVID-19 co-morbidities, will identify beneficial electro-chemical pathways related to stress, pain and memory, for example through activation of specific neurotransmitters and neuropeptides (dopamine, endorphine, serotonin). This digital health science is young but may become highly beneficial in the absence of universal vaccines and treatments for the scale and inflammatory novelties of SARS-Cov2, its variants and mutations.

ELIGIBILITY:
Inclusion Criteria:

* hospitalization for confirmed SARS-CoV-2 infection
* moderate-to-severe COVID-19 as demonstrated by the presence of typical lesions on the chest CT scan
* increased risk for cytokine storm (CRP>46mg/L, ferritin>250ng/mL)

Exclusion Criteria:

* critically ill patients upon presentation requiring direct admission to ICU

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 83 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2022-03-31 (Actual)

PRIMARY OUTCOMES:
Rate of ICU admission | From the date of study enrollment until the documented date of transfer to Intensive Care Unit (ICU), assessed up until 60 days post hospital admission

SECONDARY OUTCOMES:
Need for non-invasive ventilatory support | From the date of study enrollment until hospital discharge or death, assessed up to 60 days post hospital admission
Need for mechanical ventilation | From the date of study enrollment until hospital discharge or death, assessed up to 60 days post hospital admission
Mortality rate | From the date of study enrollment until hospital discharge, assessed up to 60 days post hospital admission

CONTACTS AND LOCATIONS:
Overall Officials: Cristian Oancea, University Professor, MD, PhD, Principal Investigator — University of Medicine and Pharmacy "Victor Babes" Timisoara
Locations (1):
- Infectious Diseases and Pulmonology Clinical Hospital Timisoara, Timișoara, Timiș County, Romania

IPD SHARING:
Plan to Share IPD: Undecided